CLINICAL TRIAL: NCT01227200
Title: The Efficiency of DYPIRON and TRAMADOL in Addition to Local Anesthesia Prior to Incision and Drainage Procedure in Peritonsillar Abscess
Brief Title: The Effect of Adding Pain Relievers to Local Anesthesia Before Preforming Drainage in Peritonsillar Abscess
Acronym: pta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: orolaryngology department, HaEmek MC
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: emc100061ctil
Record Dates: First submitted 2010-10-21; First posted 2010-10-25 (Estimated); Last update posted 2010-10-25 (Estimated); Status verified 2010-10

CONDITIONS: Peritonsillar Abscess
MeSH Terms: conditions — Peritonsillar Abscess | interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: dypiron, tramadol — dypiron 4 ML, tramadol 50 mg flashtab

SUMMARY:
The purpose of this study is to find if adding oral pain relievers as DYPIRON and TRAMADOL in addition to the local anesthesia injection, can help reducing the pain intensity in patients who diagnosed as Suffering from peritonsillar abscess (PTA)and treated by incision and drainage .

DETAILED DESCRIPTION:
Control group: the patient will get local anesthesia injection with Lidocain. After 5 minutes- the DR will preform the incision and drainage of the abscess.

Then the patient will be asked by the vas score, the the pain intensity that he feels.

Intervention group:the patient will get dypiron 4 ml and tramadol 50 mg. after 40 minutes,the patient will get local anesthesia injection with Lidocain. After 5 minutes- the DR will preform the incision and drainage of the abscess.then the patient will be asked by the vas score, the the pain intensity that he feels.

ELIGIBILITY:
Inclusion Criteria:patients with PTA in ages 18-65, who agreed to join the research -

Exclusion Criteria:cave to dypiron and/or tramadol, pregnant women, mental illness,soldiers.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2011-11; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
the vas scale | 40 min after giving the oral drugs

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - otolaryngology department, HaEmek mc, Afula
  - Otolaryngology department, HaEmek MC, Afula